CLINICAL TRIAL: NCT03839173
Title: Growth and Nutritional Status of Very Low Birth Weight Infants Fed a High Protein Exclusive Human Milk Diet
Acronym: MedolacHMF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Augusta University (Other)
Collaborators: Neolac Inc dba Medolac Laboratories (Industry)
Responsible Party: Principal Investigator, Amy Gates, Registered Dietitian and Pediatric Nutrition Specialist, Augusta University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1147989-3
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Premature Infant; Breast Milk Expression
Keywords: premature infant; breast milk; breastmilk; human milk; human milk fortifier
MeSH Terms: conditions — Premature Birth; Breast Milk Expression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrospective Chart Review (No Intervention): Retrospective Chart Review for historical controls. Historic controls fed cow's milk fortifier
- Prospective (Experimental): All neonates with birth weights ranging from 750-1500 grams and gestational ages 23-33 weeks admitted to the NICU at Augusta University within 24 hours of life will be eligible for screening within 72 hours of admission and upon parent's or legal guardian's consent.
  Infants will be fed a human milk fortifier made with donor human milk. Data will be compared with historic control data.
  Interventions: Other: Human milk based human milk fortifier

INTERVENTIONS:
Other: Human milk based human milk fortifier — A human milk fortifier with added minerals made from donor human milk
  Arms: Prospective

SUMMARY:
The purpose of this two-arm investigation is to determine if growth patterns of very low birth weight infants (VLBW) (birth weight 750-1500 grams) fed human milk (maternal or donor) supplemented with a human milk-based fortifier grow according to established guidelines and maintain adequate micronutrient levels.

DETAILED DESCRIPTION:
To achieve this goal, the investigators will prospectively analyze the growth and micronutrient status of VLBW infants who are fed human milk (maternal or donor) supplemented with a human-milk-based fortifier with increased protein (Medolac® Human Milk Fortifier). In addition, the investigators will compare the findings to retrospectively collected data for growth rates and micronutrient status of infants who received human milk fortified with cow's milk -based fortifier (Enfamil® Hydrolyzed Liquid Human Milk Fortifier). The investigators hypothesize that a human milk-based fortifier with increased protein will support growth at recommended levels (weight gain of 12-18 g/kg/day, head circumference 0.75-1.0 cm/week, length 0.8-1.1 cm/week)[1-3] and prevent micronutrient deficiency in the VLBW infant

Aim 1: To determine if VLBW infants fed human milk, maternal or donor, supplemented with a human milk-based fortifier with increased protein grow at recommended levels for weight, length, and head circumference. To achieve this aim, Z-scores for weight, length, and head circumference will be tracked. Measurements will be taken at birth and then weekly until 36 weeks post-menstrual age (PMA) or discharge from the neonatal intensive care unit (NICU), whichever comes first. Aim 2: To measure nutritional status in VLBW premature infants fed human milk supplemented with a human milk-based fortifier with increased protein. To achieve this aim, serum magnesium, potassium, chloride, blood urea nitrogen (BUN), creatinine, sodium, calcium, phosphorus, CO2, Vitamin D 1, 25 (OH) 2D, parathyroid hormone (PTH), alkaline phosphatase, hemoglobin, hematocrit will be measured within 24 hours of reaching full enteral feedings and repeated seven days later, and then every fourteen days until 36 weeks PMA or discharge, whichever comes first. Urine magnesium and sodium will be measured on the same schedule.

Aim 3: To compare growth rates and nutritional status of VLBW infants fed human milk fortified with a human milk-based fortifier to growth rates and nutritional status of those fed human milk fortified with a cow's milk-based fortifier.

ELIGIBILITY:
Inclusion Criteria:

1. Birth weight 750-1800 grams
2. Admitted to AU NICU within 24 hours of life
3. Estimated gestational age (EGA) 23 to 33 weeks as confirmed by the Ballard score
4. Birth weight appropriate for gestational age (AGA) defined as >3rd% on a gender-specific Fenton growth curve (Fenton 2013, Calgary, Canada)
5. Enteral feedings initiated within 7 days of life
6. Breastmilk diet, maternal or donor milk

Exclusion Criteria:

1. Renal conditions affecting electrolyte metabolism and/or excretion
2. Gastro-intestinal conditions that preclude feeding or affect nutrient absorption (gastroschisis, omphalocele)
3. EGA >33 weeks or birth weight >1800 grams or EGA <23 weeks or birth weight <750 grams
4. Apgar <3 at 5 minutes
5. Grade 3 or higher intraventricular hemorrhage (IVH)
6. Intrauterine growth restriction (IUGR), as defined as <3rd% on a gender-specific Fenton growth curve
7. Congenital anomalies including congenital heart disease or other major defect requiring surgical intervention
8. Intake of cow's milk formula or fortifier before or after the initiation of the study protocol

Ages: 23 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Estimated)
Dates: Start 2019-07-25 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Return to birth weight day | birth to 30 days
  Day of life infant returns to birth weight
Growth Velocity | Weekly until 36 weeks post menstrual age or discharge
  rate of weight gain measured as g/kg/day
Mean Serum Magnesium | Every 14 days until 36 weeks post menstrual age or discharge
  Serum and urine Magnesium
Mean Serum CO2 | Every 14 days until 36 weeks post menstrual age or discharge
  Serum CO2

SECONDARY OUTCOMES:
Mean z-scores | Weekly until 36 weeks post menstrual age or discharge
  z-scores for weight, length, and head circumference
Mean serum Vitamin D, 1 25 (OH) 2D | Every 14 days until 36 weeks post menstrual age or discharge
  serum Vitamin D
Mean serum parathyroid Hormone (PTH) | Every 14 days until 36 weeks post menstrual age or discharge
  Serum PTH
Mean serum Sodium | Every 14 days until 36 weeks post menstrual age or discharge
  Serum and urine Sodium
Mean serum Blood Urea Nitrogen (BUN) | Every 14 days until 36 weeks post menstrual age or discharge
  serum BUN
Mean serum Calcium | Every 14 days until 36 weeks post menstrual age or discharge
  serum Calcium
Mean serum Phosphorus | Every 14 days until 36 weeks post menstrual age or discharge
  serum Phosphorus
Mean serum Alkaline Phosphatase | Every 14 days until 36 weeks post menstrual age or discharge
  serum Alkaline Phosphatase
Mean serum Hemoglobin | Every 14 days until 36 weeks post menstrual age or discharge
  serum Hemoglobin
Mean serum Potassium | Every 14 days until 36 weeks post menstrual age or discharge
  serum and urine Potassium
Mean serum Hematocrit | Every 14 days until 36 weeks post menstrual age or discharge
  serum Hematocrit

CONTACTS AND LOCATIONS:
Overall Officials: Amy Gates, RD, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ehrenkranz RA, Dusick AM, Vohr BR, Wright LL, Wrage LA, Poole WK. Growth in the neonatal intensive care unit influences neurodevelopmental and growth outcomes of extremely low birth weight infants. Pediatrics. 2006 Apr;117(4):1253-61. doi: 10.1542/peds.2005-1368. PMID 16585322
- [Background] Fenton TR, Kim JH. A systematic review and meta-analysis to revise the Fenton growth chart for preterm infants. BMC Pediatr. 2013 Apr 20;13:59. doi: 10.1186/1471-2431-13-59. PMID 23601190
- [Background] Section on Breastfeeding. Breastfeeding and the use of human milk. Pediatrics. 2012 Mar;129(3):e827-41. doi: 10.1542/peds.2011-3552. Epub 2012 Feb 27. PMID 22371471
- [Background] Koletsko B PB, Uauy R. Nutritional Care of Preterm Infants. Basel, Switzerland: Karger, 2014.
- [Background] Kim JH, Chan G, Schanler R, Groh-Wargo S, Bloom B, Dimmit R, Williams L, Baggs G, Barrett-Reis B. Growth and Tolerance of Preterm Infants Fed a New Extensively Hydrolyzed Liquid Human Milk Fortifier. J Pediatr Gastroenterol Nutr. 2015 Dec;61(6):665-71. doi: 10.1097/MPG.0000000000001010. PMID 26488118
- [Background] Moya F, Sisk PM, Walsh KR, Berseth CL. A new liquid human milk fortifier and linear growth in preterm infants. Pediatrics. 2012 Oct;130(4):e928-35. doi: 10.1542/peds.2011-3120. Epub 2012 Sep 17. PMID 22987877
- [Background] Sullivan S, Schanler RJ, Kim JH, Patel AL, Trawoger R, Kiechl-Kohlendorfer U, Chan GM, Blanco CL, Abrams S, Cotten CM, Laroia N, Ehrenkranz RA, Dudell G, Cristofalo EA, Meier P, Lee ML, Rechtman DJ, Lucas A. An exclusively human milk-based diet is associated with a lower rate of necrotizing enterocolitis than a diet of human milk and bovine milk-based products. J Pediatr. 2010 Apr;156(4):562-7.e1. doi: 10.1016/j.jpeds.2009.10.040. Epub 2009 Dec 29. PMID 20036378
- [Background] Gates A BJ. [Neonatal Outcomes Augusta Univeristy NICU] Unpublished raw data. Augusta 2017.
- [Background] Stoll BJ, Hansen NI, Bell EF, Shankaran S, Laptook AR, Walsh MC, Hale EC, Newman NS, Schibler K, Carlo WA, Kennedy KA, Poindexter BB, Finer NN, Ehrenkranz RA, Duara S, Sanchez PJ, O'Shea TM, Goldberg RN, Van Meurs KP, Faix RG, Phelps DL, Frantz ID 3rd, Watterberg KL, Saha S, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Neonatal outcomes of extremely preterm infants from the NICHD Neonatal Research Network. Pediatrics. 2010 Sep;126(3):443-56. doi: 10.1542/peds.2009-2959. Epub 2010 Aug 23. PMID 20732945
- [Background] Thoene M, Hanson C, Lyden E, Dugick L, Ruybal L, Anderson-Berry A. Comparison of the effect of two human milk fortifiers on clinical outcomes in premature infants. Nutrients. 2014 Jan 3;6(1):261-75. doi: 10.3390/nu6010261. PMID 24394538
- [Background] Kumar N, Monga R, Sampath V, Ehrhart B. Prospective Comparison of Enfamil and Similac Liquid Human Milk Fortifier on Clinical Outcomes in Premature Infants. Am J Perinatol. 2017 Dec;34(14):1411-1416. doi: 10.1055/s-0037-1603940. Epub 2017 Jun 21. No abstract available. PMID 28637062
- [Background] Cristofalo EA, Schanler RJ, Blanco CL, Sullivan S, Trawoeger R, Kiechl-Kohlendorfer U, Dudell G, Rechtman DJ, Lee ML, Lucas A, Abrams S. Randomized trial of exclusive human milk versus preterm formula diets in extremely premature infants. J Pediatr. 2013 Dec;163(6):1592-1595.e1. doi: 10.1016/j.jpeds.2013.07.011. Epub 2013 Aug 20. PMID 23968744
- [Background] Gross SJ. Growth and biochemical response of preterm infants fed human milk or modified infant formula. N Engl J Med. 1983 Feb 3;308(5):237-41. doi: 10.1056/NEJM198302033080501. PMID 6848932
- [Background] Agostoni C, Buonocore G, Carnielli VP, De Curtis M, Darmaun D, Decsi T, Domellof M, Embleton ND, Fusch C, Genzel-Boroviczeny O, Goulet O, Kalhan SC, Kolacek S, Koletzko B, Lapillonne A, Mihatsch W, Moreno L, Neu J, Poindexter B, Puntis J, Putet G, Rigo J, Riskin A, Salle B, Sauer P, Shamir R, Szajewska H, Thureen P, Turck D, van Goudoever JB, Ziegler EE; ESPGHAN Committee on Nutrition. Enteral nutrient supply for preterm infants: commentary from the European Society of Paediatric Gastroenterology, Hepatology and Nutrition Committee on Nutrition. J Pediatr Gastroenterol Nutr. 2010 Jan;50(1):85-91. doi: 10.1097/MPG.0b013e3181adaee0. PMID 19881390
- [Background] Ong KK, Kennedy K, Castaneda-Gutierrez E, Forsyth S, Godfrey KM, Koletzko B, Latulippe ME, Ozanne SE, Rueda R, Schoemaker MH, van der Beek EM, van Buuren S, Fewtrell M. Postnatal growth in preterm infants and later health outcomes: a systematic review. Acta Paediatr. 2015 Oct;104(10):974-86. doi: 10.1111/apa.13128. PMID 26179961
- [Background] Ghandehari H, Lee ML, Rechtman DJ; H2MF Study Group. An exclusive human milk-based diet in extremely premature infants reduces the probability of remaining on total parenteral nutrition: a reanalysis of the data. BMC Res Notes. 2012 Apr 25;5:188. doi: 10.1186/1756-0500-5-188. PMID 22534258
- [Background] Food and Drug Administration, HHS. Current good manufacturing practices, quality control procedures, quality factors, notification requirements, and records and reports, for infant formula. Final rule. Fed Regist. 2014 Jun 10;79(111):33057-72. PMID 24922980